CLINICAL TRIAL: NCT04444700
Title: Utilização da Enoxaparina em Dose Anticoagulante em Pacientes Hospitalizados Com síndrome respiratória Aguda Grave Por COVID-19
Brief Title: A Pragmatic Randomized Controlled Trial of Therapeutic Anticoagulation Versus Standard Care as a Rapid Response to (SARS-CoV-2) COVID-19 Pandemic
Acronym: RAPID-BRAZIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Unity Health Toronto (Other); University of Vermont Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 33109220.7.0000.0068
Record Dates: First submitted 2020-06-22; First posted 2020-06-23 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID; Coronavirus Infection; Severe Acute Respiratory Syndrome; Thromboembolism, Venous; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; Venous Thromboembolism; Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm, parallel, pragmatic, multi-centre, open-label randomized controlled trial to determine the effect of therapeutic anticoagulation on the composite outcome of ICU admission, mechanical ventilation and/or death in hospitalized patients with COVID-19.
Masking Description: None (Open Label) Blinding of participants, clinical research staff, and clinicians is not possible due to the nature of the intervention. However, the biostatisticians will be blinded at the data analysis phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic anticoagulation (Experimental): Therapeutic anticoagulation with LMWH or UFH (high dose nomogram). The choice of LMWH versus UFH will be at the clinician's discretion and dependent on local institutional supply. Therapeutic anticoagulation will be administered until discharged from hospital, 28 days or death. If the patient is admitted to the ICU or requiring ventilatory support, we recommend continuation of the allocated treatment as long as the treating physician is in agreement.
  Interventions: Drug: Therapeutic anticoagulation
- Standard care (No Intervention): Administration of LMWH, UFH or fondaparinux at thromboprophylactic doses for acutely ill hospitalized medical patients, in the absence of contraindication, is considered standard care.

INTERVENTIONS:
Drug: Therapeutic anticoagulation — The choice of low molecular weight heparin (LMWH) versus unfractionated heparin (UFH) will be at the clinician's discretion. LMWH options include: Tinzaparin, Enoxaparin or Dalteparin. UFH will be administered using a weight-based nomogram with titration according to center-specific institutional protocol.
  Arms: Therapeutic anticoagulation

SUMMARY:
Coagulopathy of COVID-19 afflicts approximately 20% of patients with severe COVID-19 and is associated with need for critical care and death. COVID-19 coagulopathy is characterized by elevated D-dimer, an indicator of fibrin formation and clot lysis, and a mildly prolonged prothrombin time, suggestive of coagulation consumption. To date, it seems that COVID-19 coagulopathy manifests with thromboembolism, thus anticoagulation may be of benefit. We propose to conduct a parallel pragmatic multi-centre open-label randomized controlled trial to determine the effect of therapeutic anticoagulation compared to standard care in hospitalized patients admitted for COVID-19 with an elevated D-dimer.

DETAILED DESCRIPTION:
2-arm, parallel, pragmatic, multi-centre, open-label randomized controlled trial to determine the effect of therapeutic anticoagulation, with low molecular weight heparin or unfractionated heparin (high dose nomogram), compared to standard care in hospitalized patients with COVID-19 and an elevated D-dimer on the composite outcome of intensive care unit (ICU) admission, non-invasive positive pressure ventilation, invasive mechanical ventilation or death at 28 days. Eligible participants will be randomized to one of two treatment regimens, receiving either therapeutic anticoagulation or standard care until discharged from hospital, death or day 28.

The primary composite outcome of ICU admission, non-invasive positive pressure ventilation, invasive mechanical ventilation, or all-cause death up to 28 days.

Key secondary outcomes between study arms up to day 28 include:

1. All-cause death
2. Composite outcome of ICU admission or all-cause death
3. Composite outcome of mechanical ventilation or all-cause death
4. Major bleeding as defined by the ISTH Scientific and Standardization Committee (ISTH-SSC) recommendation
5. Number of participants who received red blood cell transfusion (≥1 unit)
6. Number of participants with transfusion of platelets, frozen plasma, prothrombin complex concentrate, cryoprecipitate and/or fibrinogen concentrate
7. Renal replacement therapy;
8. Number of hospital-free days alive
9. Number of ICU-free days alive
10. Number of ventilator-free days alive
11. Number of organ support-free days alive
12. Number of participants with venous thromboembolism
13. Number of participants with arterial thromboembolism
14. Number of participants with heparin induced thrombocytopenia
15. Changes in D-dimer up to day 3

The treatment arm is therapeutic anticoagulation with low molecular weight heparin (LMWH) or unfractionated heparin (UFH, high dose nomogram). The choice of LMWH versus UFH will be at the clinician's discretion. LMWH options include: Tinzaparin, Enoxaparin, or Dalteparin. UFH will be administered using a weight-based nomogram with titration according to the center-specific protocol. Therapeutic anticoagulation will be administered until discharged from hospital, 28 days or death. If the patient is admitted to the ICU or requiring ventilatory support, we recommend continuation of the allocated treatment as long as the treating physician is in agreement. The standard care arm is the administration of LMWH, UFH or fondaparinux at thromboprophylactic doses in the absence of contraindication.

No study specific bloodwork will be ordered aside from a single D-dimer test (if not collected through standard of care) up to and including day 3 after randomization for all participants in both study arms. In those on the active treatment arm who are receiving UFH, the aPTT or UFH anti-Xa will be drawn according to local institutional UFH nomogram protocol guidance. All laboratory results will be collected from standard of care from admission to hospital discharge, death or 28 days, where available. An optional biobanking component will collect blood at baseline and 2 follow up time points.

This study will immediately impact the clinical care of patients with severe COVID-19 internationally, whether the findings are positive or negative, as COVID-19 coagulopathy is a highly prevalent complication of severe COVID-19 and may precede the respiratory manifestations that characterize it.

ELIGIBILITY:
The inclusion criteria are:

1. laboratory confirmed diagnosis of SARS-CoV-2 via reverse transcriptase polymerase chain reaction as per the World Health Organization protocol or by nucleic acid based isothermal amplification.Positive test prior to hospital admission OR within first 5 days (i.e. 120 hours) after hospital admission;
2. admitted to hospital for COVID-19;
3. one D-dimer value above ULN (5 days (i.e. 120 hours) of hospital admission) and either: a) D-Dimer ≥2 times ULN; or b) D-dimer above ULN and oxygen saturation ≤ 93% on room air;
4. ≥18 years of age;
5. informed consent from the patient (or legally authorized substitute decision maker).

The exclusion criteria are:

1. pregnancy;
2. hemoglobin <80 g/L in the last 72 hours;
3. platelet count <50 x 10^9/L in the last 72 hours;
4. known fibrinogen <1.5 g/L (if testing deemed clinically indicated by the treating physician prior to the initiation of anticoagulation);
5. known INR >1.8 (if testing deemed clinically indicated by the treating physician prior to the initiation of anticoagulation);
6. patient already on intermediate dosing of LMWH that cannot be changed (determination of what constitutes an intermediate dose is to be at the discretion of the treating clinician taking the local institutional thromboprophylaxis protocol for high risk patients into consideration);
7. patient already on therapeutic anticoagulation at the time of screening (low or high dose nomogram UFH, LMWH, warfarin, direct oral anticoagulant (any dose of dabigatran, apixaban, rivaroxaban, edoxaban);
8. patient on dual antiplatelet therapy, when one of the agents cannot be stopped safely;
9. known bleeding within the last 30 days requiring emergency room presentation or hospitalization;
10. known history of a bleeding disorder of an inherited or active acquired bleeding disorder;
11. known history of heparin-induced thrombocytopenia;
12. known allergy to UFH or LMWH;
13. admitted to the intensive care unit at the time of screening;
14. treated with non-invasive positive pressure ventilation or invasive mechanical ventilation at the time of screening (of note: high flow oxygen delivery via nasal cannula is acceptable and is not an exclusion criterion).
15. imminent death according to the judgement of the most responsible physician
16. enrollment in another clinical trial of antithrombotic therapy involving pre-intensive care unit hospitalized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Composite outcome of ICU admission (yes/no), non-invasive positive pressure ventilation (yes/no), invasive mechanical ventilation (yes/no), or all-cause death (yes/no) up to 28 days. | up to 28 days
  Composite outcome of ICU admission (yes/no), non-invasive positive pressure ventilation (yes/no), invasive mechanical ventilation (yes/no), or all-cause death (yes/no) up to 28 days.

SECONDARY OUTCOMES:
All-cause death | Up to 28 days
  All-cause death
Composite outcome of ICU admission or all-cause death | Up to 28 days
  Composite outcome of ICU admission or all-cause death
Composite outcome of mechanical ventilation or all-cause death | Up to 28 days
  Composite outcome of mechanical ventilation or all-cause death
Major bleeding | Up to 28 days
  Major bleeding as defined by the ISTH Scientific and Standardization Committee (ISTH-SSC) recommendation
Red blood cell transfusion | Up to 28 days
  Red Blood Cell transfusion (greater than or equal to 1 unit)
Transfusion of platelets, frozen plasma, prothrombin complex concentrate, cryoprecipiate and/or fibrinogen concentrate | Up to 28 days
  Transfusion of platelets, frozen plasma, prothrombin complex concentrate, cryoprecipiate and/or fibrinogen concentrate
Renal replacement therapy | Up to 28 days
  Renal replacement therapy defined as continuous renal replacement therapy or intermittent hemodialysis
Hospital-free days alive up to day 28 | Up to 28 days
  Hospital-free days alive up to day 28
ICU-free days alive up to day 28 | Up to 28 days
  ICU-free days alive up to day 28
Ventilator-free days alive up to day 28 | Up to 28 days
  Ventilator-free days alive up to day 28
Organ support-free days alive up to day 28 | Up to 28 days
  Organ support-free days alive up to day 28
Venous thromboembolism | Up to 28 days
  Venous thromboembolism
Arterial thromboembolism | Up to 28 days
  Arterial thromboembolism
Heparin induced thrombocytopenia | Up to 28 days
  Heparin induced thrombocytopenia
Changes in D-dimer up to day 3 | Up to day 3
  D-dimer

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juni, MD, FESC, Principal Investigator — St Michael's Hospital, Li Ka Shing Knowledge Institute, University of Toronto; Elnara M Negri, MD, PhD, Principal Investigator — Laboratório de Investigação Médica da FMUSP; Heraldo P de Souza, MD, PhD, Principal Investigator — Disciplina de Emergências Clínicas, Hospital das Clínicas da FMUSP; Hassan Rahhal, MD, Principal Investigator — Disciplina de Emergências Clínicas, Hospital das Clínicas da FMUSP
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sholzberg M, Tang GH, Rahhal H, AlHamzah M, Kreuziger LB, Ni Ainle F, Alomran F, Alayed K, Alsheef M, AlSumait F, Pompilio CE, Sperlich C, Tangri S, Tang T, Jaksa P, Suryanarayan D, Almarshoodi M, Castellucci L, James PD, Lillicrap D, Carrier M, Beckett A, Colovos C, Jayakar J, Arsenault MP, Wu C, Doyon K, Andreou ER, Dounaevskaia V, Tseng EK, Lim G, Fralick M, Middeldorp S, Lee AYY, Zuo F, da Costa BR, Thorpe KE, Negri EM, Cushman M, Juni P; RAPID Trial investigators. Heparin for Moderately Ill Patients with Covid-19. medRxiv [Preprint]. 2021 Jul 12:2021.07.08.21259351. doi: 10.1101/2021.07.08.21259351. PMID 34268513